CLINICAL TRIAL: NCT06590545
Title: Anti-CD 19 CAR-T Cell Therapy in Patients with ANCA Vasculitis: a Two-stage Interventional, Prospective, Open-label, Phase I/II Trial in Patients with Active, Treatment Refractory, ANCA-IgG-positive Vasculitis
Brief Title: Anti-CD 19 CAR-T Cell Therapy in Patients with ANCA Vasculitis
Acronym: IDEAL
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: David Simon (Other)
Collaborators: Kyverna Therapeutics (Industry)
Responsible Party: Sponsor-Investigator, David Simon, Principal Investigator, Head of the Clinical Trial Unit, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CCM-RNT-202402; 2024-517303-36-00 (EU CTIS Number)
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: ANCA-IgG-positive ANCA Associated Vasculitis
Keywords: ANCA; CAR-T-Cell; Vasculitis; Seroconversion; anti-CD19
MeSH Terms: conditions — Vasculitis; HIV Seropositivity

STUDY DESIGN:
Intervention Model Description: this is a two-stage interventional, prospective, open-label study. This study has one treatment arm (open-label KYV101), but sequential treatment (two groups). Second group of participants are assigned to receive interventions based on the achievement of the previous milestone (28 days after treatment of the third patient of group 1). A data safety monitoring board (DSMB) will decide whether to proceed to phase II ≥ 28 days after treatment of the third subject.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- KYV-101, anti-CD19 CAR T-cell immunotherapy. (Experimental): A dosage of 1x10^8 KYV-101 CAR+ T cells will be administered intravenously as a single infusion.
  Interventions: Drug: KYV-101, an autologous fully-human anti-CD19 CAR T-cell immunotherapy

INTERVENTIONS:
Drug: KYV-101, an autologous fully-human anti-CD19 CAR T-cell immunotherapy — A dosage of 1x10^8 KYV-101 CAR+ T cells will be administered intravenously as a single infusion.

SUMMARY:
The goal of this phase I/II clinical trial is to investigate anti-CD 19 chimeric antigen receptor T cell (CAR-T cell) therapy in patients with antineutrophil cytoplasmic antibodies (ANCA) immunoglobulin (IgG) positive ANCA associated vasculitis (AAV).

The main questions it aims to answer are:

* To assess the safety of anti-CD19 CAR-T cell therapy in subjects with active, treatment refractory, ANCA-IgG-positive AAV
* To assess the clinical efficacy of anti-CD19 CAR-T cell therapy in subjects with active, treatment refractory ANCA-IgG-positive AAV
* To assess the ANCA seroconversion rate in subjects with active, treatment refractory ANCA-IgG-positive AAV

Participants will receive a single dose of KYV-101 i.v., an autologous fully-human anti-CD19 CAR-T cell immunotherapy. Follow-up time is 52 weeks with regular visits at the site.

DETAILED DESCRIPTION:
This study aims to investigate the use of KYV101 (a fully human anti-CD19 CAR T cell therapy) in ANCA-IgG-positive AAV patients who are refractory to previous treatments. This study is designed to determine (i) the safety of this B-cell targeted therapy, (ii) the clinical efficacy, (iii) the impact on the immunological status of the patient and in particular on ANCA positivity, and (iv) the ability to induce long-term (deep) clinical and molecular remission and drug-free survival.

The investigational product (IMP), KYV-101, is an autologous fully-human anti-CD19 CAR T-cell immunotherapy. Before IMP infusion, patients will receive a premedication of 4 mg Dimetindenmaleat iv or equivalent antihistamine and 1000 mg oral acetaminophene. Prophylactic doses of acyclovir of 400mg 2x daily as well as cotrimoxazole 960mg 3x weekly will be administered orally following CAR T cell infusion until week 24. Tocilizumab 8mg/kg will be administered intravenously when required for treatment of IMP-related cytokine release syndrome. Dexamethasone as needed will be administered intravenously when required for treatment of neurological adverse event (ICANS).

Follow-up time is 52 weeks with regular visits at the site.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign an informed consent form
* Male or female, age ≥ 18 and ≤ 75 years at ti me of consent
* Able to adhere to the study visits and protocol
* Fulfilment of
* EITHER both of the following

  * 2022 ACR-EULAR classification criteria for granulomatosis with polyangiitis (GPA)
  * detectable anti-PR3 antibodies (≥ 20 AU/ml in CLIA) at screening
* OR both of the following

  * 2022 ACR/EULAR classification criteria for microscopic polyangiitis (MPA)
  * detectable anti-MPO antibodies (≥ 10 AU/ml in CLIA) at screening
* Active disease, defined as Clinical activity (BVAS ≥ 3) at screening
* Insufficient response or intolerance/contraindication to glucocorticoids and to at least one of the following treatments: rituximab, mycophenolate mofetil, azathioprine, methotrexate, cyclophosphamide, avacopan. Insufficient response is defined as having disease activity based on the definition explained in the previous bullet point
* Male subjects unless surgically sterile, must agree to use two acceptable methods for contraception (e.g. spermicide and condom) during the trial and refrain from fathering a child starting from the time of signing the Informed Consent Form (ICF) until 12 months after dosing of the IMP
* Females of childbearing potential (FCBP) must have a negative urine pregnancy test at screening and must agree to use a highly effective contraceptive method (Pearl index less than 1) starting from the time of signing the ICF and for 12 months after dosing of the IMP
* Updated vaccination record according to the STIKO recommendations for immuno-compromised patients

Exclusion Criteria:

* ANC less than 500/µl, ALC less than 100/µl or hemoglobin less than 8g/dl, absolute CD3+T cell count less than 100/µl at screening
* Severely impaired renal (eGFR ≤ 30 ml/min/m2), liver (Child Pugh C), or heart or pulmonary (NYHA IV, blood oxygenation less than 92%) function
* Clinically relevant rapidly progressive glomerulonephritis or pulmonary alveolar hemorrhage
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
* Prior treatment with anti-CD19 antibody therapy, adoptive T cell therapy or any prior gene therapy product (e.g. CAR T cell therapy)
* History of bone marrow/ hematopoietic stem cell or solid organ transplantation
* Any concomitant severe active infection, e.g. HIV, hepatitis B or C, SARS-CoV-2 (COVID-19), or active tuberculosis as defined by a positive Quantiferon TB-test. If presence of latent tuberculosis is established then treatment according to local guide-lines must have been initiated prior to enrollment
* Pregnant or lactating females
* Females who are intending to conceive during the study
* Known hypersensitivity to any drug components
* Malignancy in the last 5 years before screening (except adequately treated basal or squamous cell skin cancer)
* Requirement for immunization with live vaccine during the study period or within 14 days preceding leukapheresis,
* Subjects who are younger than 18 years or are incapable to understand the aim, importance and consequences of the study and to give legal informed consent (accord-ing to § 40 Abs. 4 and § 41 Abs. 2 and Abs. 3 AMG),
* Have a history of alcohol or substance abuse within the preceding 6 months that, in the opinion of the Investigator, may increase the risks associated with study participa-tion or study agent administration, or may interfere with interpretation of results,
* Subjects who possibly are dependent on the Sponsor, the Principal Investigator or Investigator (e.g. family members).
* Subjects who are institutionalized by order of court or public authority,
* Subjects participating in another clinical trial with an investigational medicinal product or medical device (3 months before this trial).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — all
Enrollment: 8 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
number of subjects experiencing a cytokine release syndrome | Screening up to week 4
  The primary safety outcome in Phase I variable will be measured as the number of subjects experiencing a cytokine release syndrome (CRS) or an immune cell-associated neurotoxicity syndrome (ICANS) as well as adverse events (AE) and serious adverse events (SAE) due to investigational medical product (IMP) within the first 4 weeks.
antineutrophil cytoplasmic antibodies (ANCA) seroconversion rate | week 24
  The primary efficacy outcome variable of Phase II will be the antineutrophil cytoplasmic antibodies (ANCA) seroconversion rate in subjects with active, treatment refractory ANCA-IgG-positive AAV at week 24.
adverse events and serious adverse events due to investigational medical product | up to 52 weeks
  The primary safety outcome variable of Phase II will be measured as adverse events (AE) and serious adverse events (SAE) due to investigational medical product (IMP) throughout the whole study.

SECONDARY OUTCOMES:
immunoglobulin IgG | up to week 52
  Change in total IgG immunoglobulins over time
immunoglobulin IgG subclasses | up to week 52
  Change in total IgG subclasses mmunoglobulins over time
immunoglobulin IgA | up to week 52
  Change in total IgA immunoglobulins over time
immunoglobulin IgM | up to week 52
  Change in total IgM immunoglobulins over time
Change in PR3 | up to week 52
  Change in PR3 specific plasmablasts and B-cells
Change in MPO | up to week 52
  Change in MPO specific plasmablasts and B-cells
number of plasmablasts | up to week 52
  Change in the number of plasmablasts cell over time
number of B cells | up to week 52
  Change in the number of pB cells numbers over time
number of T cells | up to week 52
  Change in the number T cells numbers over time
relapse/flare | up to 52 weeks
  Time to relapse/flare
time without immunosuppression | up to 52 weeks
  Survival time without immunosuppression
Vasculitis Damage Index | up to 52 weeks
  Change of Vasculitis Damage Index (VDI) compared to baseline
Flares | up to 52 weeks
  Number of flares
Birmingham Vasculitis Activity Score | up to 52 weeks
  Change in Birmingham Vasculitis Activity Score (BVAS) compared to baseline
B cell depletion | up to 52 weeks
  Duration of B cell depletion in the peripheral blood
persistence of CAR T cells | up to 52 weeks
  Duration of persistence of CAR T cells in the peripheral blood
Change in anti-PR3 antibodies | up to 52 weeks
  Change in anti-PR3 antibodies over time (GPA)
anti-MPO antibodies | up to 52 weeks
  Change in anti-MPO antibodies over time
anti-MPO antibodies | up to week 52
  Percentage of subjects with normal anti-MPO antibodies (less than 10 AU/ml)
normal anti-PR3 antibodies | up to 52 weeks
  Percentage of subjects with normal anti-PR3 antibodies (less than 20 AU/ml in CLIA)
EULAR sustained remission criteria | up to week 52
  Percentage of patients who reach European Alliance of Associations for Rheumatology (EULAR) sustained remission criteria (absence of typical signs, symptoms, or other features of active ANCA associated vasculitis)
reach EULAR response criteria | up to 52 weeks
  Percentage of patients who reach European Alliance of Associations for Rheumatology (EULAR) response criteria (≥ 50% reduction of Birmingham Vasculitis Activity Score (BVAS) compared to baseline
number of CAR-T cells | up to 52 weeks
  number of CAR-T cells in the patient over time

IPD SHARING:
Plan to Share IPD: No
results will be published anonymized and summarized

REFERENCES:
- [Background] Hellmich B, Sanchez-Alamo B, Schirmer JH, Berti A, Blockmans D, Cid MC, Holle JU, Hollinger N, Karadag O, Kronbichler A, Little MA, Luqmani RA, Mahr A, Merkel PA, Mohammad AJ, Monti S, Mukhtyar CB, Musial J, Price-Kuehne F, Segelmark M, Teng YKO, Terrier B, Tomasson G, Vaglio A, Vassilopoulos D, Verhoeven P, Jayne D. EULAR recommendations for the management of ANCA-associated vasculitis: 2022 update. Ann Rheum Dis. 2024 Jan 2;83(1):30-47. doi: 10.1136/ard-2022-223764. PMID 36927642
- [Background] Han WK, Choi HK, Roth RM, McCluskey RT, Niles JL. Serial ANCA titers: useful tool for prevention of relapses in ANCA-associated vasculitis. Kidney Int. 2003 Mar;63(3):1079-85. doi: 10.1046/j.1523-1755.2003.00821.x. PMID 12631091
- [Background] Muller F, Taubmann J, Bucci L, Wilhelm A, Bergmann C, Volkl S, Aigner M, Rothe T, Minopoulou I, Tur C, Knitza J, Kharboutli S, Kretschmann S, Vasova I, Spoerl S, Reimann H, Munoz L, Gerlach RG, Schafer S, Grieshaber-Bouyer R, Korganow AS, Farge-Bancel D, Mougiakakos D, Bozec A, Winkler T, Kronke G, Mackensen A, Schett G. CD19 CAR T-Cell Therapy in Autoimmune Disease - A Case Series with Follow-up. N Engl J Med. 2024 Feb 22;390(8):687-700. doi: 10.1056/NEJMoa2308917. PMID 38381673
- [Background] Schett G, Mackensen A, Mougiakakos D. CAR T-cell therapy in autoimmune diseases. Lancet. 2023 Nov 25;402(10416):2034-2044. doi: 10.1016/S0140-6736(23)01126-1. Epub 2023 Sep 22. PMID 37748491
- [Background] Mackensen A, Muller F, Mougiakakos D, Boltz S, Wilhelm A, Aigner M, Volkl S, Simon D, Kleyer A, Munoz L, Kretschmann S, Kharboutli S, Gary R, Reimann H, Rosler W, Uderhardt S, Bang H, Herrmann M, Ekici AB, Buettner C, Habenicht KM, Winkler TH, Kronke G, Schett G. Anti-CD19 CAR T cell therapy for refractory systemic lupus erythematosus. Nat Med. 2022 Oct;28(10):2124-2132. doi: 10.1038/s41591-022-02017-5. Epub 2022 Sep 15. PMID 36109639
- [Background] Mougiakakos D, Kronke G, Volkl S, Kretschmann S, Aigner M, Kharboutli S, Boltz S, Manger B, Mackensen A, Schett G. CD19-Targeted CAR T Cells in Refractory Systemic Lupus Erythematosus. N Engl J Med. 2021 Aug 5;385(6):567-569. doi: 10.1056/NEJMc2107725. No abstract available. PMID 34347960
- [Background] Lodka D, Zschummel M, Bunse M, Rousselle A, Sonnemann J, Kettritz R, Hopken UE, Schreiber A. CD19-targeting CAR T cells protect from ANCA-induced acute kidney injury. Ann Rheum Dis. 2024 Mar 12;83(4):499-507. doi: 10.1136/ard-2023-224875. PMID 38182404
- [Background] Treppo E, Binutti M, Agarinis R, De Vita S, Quartuccio L. Rituximab Induction and Maintenance in ANCA-Associated Vasculitis: State of the Art and Future Perspectives. J Clin Med. 2021 Aug 24;10(17):3773. doi: 10.3390/jcm10173773. PMID 34501224
- [Background] Steinmetz OM, Velden J, Kneissler U, Marx M, Klein A, Helmchen U, Stahl RA, Panzer U. Analysis and classification of B-cell infiltrates in lupus and ANCA-associated nephritis. Kidney Int. 2008 Aug;74(4):448-57. doi: 10.1038/ki.2008.191. Epub 2008 Jun 4. PMID 18528326
- [Background] Holden NJ, Williams JM, Morgan MD, Challa A, Gordon J, Pepper RJ, Salama AD, Harper L, Savage CO. ANCA-stimulated neutrophils release BLyS and promote B cell survival: a clinically relevant cellular process. Ann Rheum Dis. 2011 Dec;70(12):2229-33. doi: 10.1136/ard.2011.153890. Epub 2011 Aug 21. PMID 21859691
- [Background] Falk RJ, Terrell RS, Charles LA, Jennette JC. Anti-neutrophil cytoplasmic autoantibodies induce neutrophils to degranulate and produce oxygen radicals in vitro. Proc Natl Acad Sci U S A. 1990 Jun;87(11):4115-9. doi: 10.1073/pnas.87.11.4115. PMID 2161532
- [Background] Kitching AR, Anders HJ, Basu N, Brouwer E, Gordon J, Jayne DR, Kullman J, Lyons PA, Merkel PA, Savage COS, Specks U, Kain R. ANCA-associated vasculitis. Nat Rev Dis Primers. 2020 Aug 27;6(1):71. doi: 10.1038/s41572-020-0204-y. PMID 32855422
- [Background] Brudno JN, Lam N, Vanasse D, Shen YW, Rose JJ, Rossi J, Xue A, Bot A, Scholler N, Mikkilineni L, Roschewski M, Dean R, Cachau R, Youkharibache P, Patel R, Hansen B, Stroncek DF, Rosenberg SA, Gress RE, Kochenderfer JN. Author Correction: Safety and feasibility of anti-CD19 CAR T cells with fully human binding domains in patients with B-cell lymphoma. Nat Med. 2020 May;26(5):803. doi: 10.1038/s41591-020-0864-x. PMID 32291416